CLINICAL TRIAL: NCT01055444
Title: An Open-Label Pilot Study Evaluating Synera® in the Treatment of Patients With Shoulder Impingement Syndrome
Brief Title: Study Evaluating Heated Lidocaine/Tetracaine Topical Patch in Treatment of Patients With Shoulder Impingement Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ZARS Pharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SC-202
Record Dates: First submitted 2010-01-21; First posted 2010-01-25 (Estimated); Last update posted 2012-03-16 (Estimated); Status verified 2012-03

CONDITIONS: Shoulder Impingement Syndrome
MeSH Terms: conditions — Shoulder Impingement Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Heated lidocaine/tetracaine topical patch (Experimental): Patients will be instructed to apply one heated lidocaine 70 mg and tetracaine 70 mg topical patch to the affected shoulder every 12 hours starting on the evening of Day 1 through the morning of Day 14 (morning and evening applications) and to remove the patch after 2-4 hours.
  Interventions: Drug: Heated lidocaine and tetracaine topical patch

INTERVENTIONS:
Drug: Heated lidocaine and tetracaine topical patch — Patients will be instructed to apply one heated lidocaine 70 mg and tetracaine 70 mg topical patch to the affected shoulder every 12 hours starting on the evening of Day 1 through the morning of Day 14 (morning and evening applications) and to remove the patch after 2-4 hours.
  Other Names: Synera

SUMMARY:
The purpose of the study is to explore the potential usefulness of a heated lidocaine 70 mg/tetracaine 70 mg topical patch for the treatment of pain associated with shoulder impingement syndrome

DETAILED DESCRIPTION:
The purpose of this single center, 2-week open-label pilot study is to explore the potential usefulness of a heated lidocaine 70 mg and tetracaine 70 mg topical patch for the treatment of pain associated with shoulder impingement syndrome. A number of efficacy variables will be employed to evaluate their utility for assessing painful responses in this population.

ELIGIBILITY:
Inclusion Criteria:

* Pain associated with shoulder impingement syndrome in a single shoulder
* Have tenderness at the attachment site of the rotator cuff tendons in the affected shoulder
* Have positive Hawkins and Neers signs

Exclusion Criteria:

* Have used any topically applied pain medication on the target treatment area within 3 days preceding the Screening/Baseline visit
* Have used any injected pain medication within 14 days preceding the Screening/Baseline visit
* Are receiving class 1 antiarrhythmic drugs (ie, tocainide, mexiletine, etc.)
* Have a history of and/or past diagnosis of severe hepatic disease

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-03; Primary Completion 2010-08 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Pain intensity | Two weeks

SECONDARY OUTCOMES:
Pain interference with activities (general, normal work, and sleep) | Two weeks

CONTACTS AND LOCATIONS:
Overall Officials: Richard Radnovich, DO, Principal Investigator
Locations (1):
- Injury Care Medical Center, Boise, Idaho, United States